CLINICAL TRIAL: NCT01028235
Title: Routine Screening for Eosinophilic Esophagitis in Patients Presenting With Dysphagia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Antonio Uniformed Services Health Education Consortium (U.S. Federal Agency)
Responsible Party: Jonathan M. Ricker, DO Gastroenterology Fellow, SAUSHEC
Other Study IDs: FWH20060112H
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-11

CONDITIONS: Dysphagia
Keywords: Eosinophilic Esophagitis
MeSH Terms: conditions — Deglutition Disorders; Eosinophilic Esophagitis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 endoscopic biopsies from 5 locations: duodenum, stomach, distal esophagus, mid esophagus and proximal esophagus
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obstructive Dysphagia: Patients who complained of dysphagia, which had an obstructive etiology for their symptoms at the time of endoscopy (ring, mass, stricture, etc)
- Non-obstructive Dysphagia: Patients whose endoscopy was normal and without any obvious etiology for their symptoms noted.

SUMMARY:
The purpose of this study is to identify the prevalence of pathologic eosinophilic esophagitis (EoE) in the cohort of adult patients who present for specialty care in the gastroenterology clinics with complaint of difficulty swallowing (dysphagia). From this, the investigators will make recommendations regarding routine screening for the diagnosis in this cohort. The prevalence of EoE in patients presenting for specialty care in the gastroenterology clinics with the complaint of dysphagia is great enough that the diagnosis should be routinely screened against in this cohort.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* complaint of dysphagia

Exclusion Criteria:

* pregnancy
* age <18
* on inhaled steroids within the last 30 days
* on systemic steroids in the last 30 days
* known diagnosis of Eosinophilic Esophagitis
* obvious obstructive etiology found at endoscopy
* increased risk of bleeding (on blood thinners or anti-platelet agents other than aspirin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients over age 18, presenting to the Gastroenterology Clinic with the complaint of dysphagia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Ricker, DO, Principal Investigator — San Antonio Uniformed Services Health Education Consortium
Locations (2):
- United States (2):
  - Wilford Hall Medical Center, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas